CLINICAL TRIAL: NCT03797677
Title: A Pilot Study to Evaluate the Use of the MN4000 for Treatment of Cystic Fibrosis (CF) and Motor Neuron Disease (MND) Patients in the Home Setting
Brief Title: MN4000 for Treatment of CF and MND Patients in the Home Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hill-Rom (Industry)
Responsible Party: Sponsor
Organization: Baxter Healthcare Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-RR2016-002
Record Dates: First submitted 2018-12-27; First posted 2019-01-09 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Cystic Fibrosis; Motor Neuron Disease; Airway Clearance Impairment
Keywords: Airway Clearance; Cystic Fibrosis; Motor Neuron Disease; Home care
MeSH Terms: conditions — Cystic Fibrosis; Motor Neuron Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Home based airway clearance with Metaneb (Experimental): Patients with CF and MND who required regular home airway clearance therapy were enrolled to use the Metaneb device in the home setting.
  The MN4000 is an airway clearance and lung expansion therapy device that has been cleared to market by the FDA as The MetaNeb® System for Homecare environment, for clearance of pulmonary secretions and for treatment or prevention of pulmonary atelectasis. It is a Class II device, cleared to market on March 17, 2016 under premarket notification 510(k) K151689 as The MetaNeb® 4 System with application for homecare environment.
  Interventions: Device: MN 4000

INTERVENTIONS:
Device: MN 4000 — Patients who required regular home airway clearance therapy were enrolled in the study and were prescribed therapy with the MN4000. Adherence to the prescribed therapy regimen and patient/caregiver satisfaction with the therapy was assessed. Pulmonary function, was assessed for each subject at baseline, after 1 month and after 3 months of home therapy. Results from the therapy period was compared to the baseline period, during which the subject received their regular airway clearance regimen. Airway Clearance Satisfaction surveys were conducted at baseline, after 1 month, and after 3 months of therapy. Results from the MN4000 therapy period were compared to the baseline period, during which the subject received their regular regimen

SUMMARY:
The study was a non-randomized open label pilot study. It was an observational design conducted at one (1) site in the US. All enrolled subjects received treatment with the MN4000.

This pilot study evaluated subject satisfaction with the therapy and adherence to the therapy during the 90-day treatment period, and also collected clinical outcome data. Outcomes were assessed before, during and after the MN4000 treatment period.

DETAILED DESCRIPTION:
The study was a non-randomized open label pilot study. It was an observational design conducted at one (1) site in the US. All enrolled subjects received treatment with the MN4000.

This pilot study evaluated subject satisfaction with the therapy and adherence to the therapy during the 90-day treatment period, and also collected clinical outcome data. Outcomes were assessed before, during and after the MN4000 treatment period. The study did not include a control group. This pilot study was designed to provide initial information that could inform decisions for future larger-scale studies.

Ten (10) patients total were enrolled from CF and NMD clinics. Eligible subjects were adult patients who were able to perform MN4000 therapy using a mouthpiece and who met all inclusion and none of the exclusion criteria.

All patients received therapy with the MN4000 following the labeled instructions for the device.

The MN4000 is an airway clearance and lung expansion therapy device that has been cleared to market by the FDA as The MetaNeb® System for Homecare environment, for clearance of pulmonary secretions and for treatment or prevention of pulmonary atelectasis. It is a Class II device, cleared to market on March 17, 2016 under premarket notification 510(k) K151689 as The MetaNeb® 4 System with application for homecare environment. It is commercially marketed as the MN4000. The device consists of a pneumatic compressor and an air pulse generator that delivers CHFO and CPEP to;

1. facilitate clearance of mucous from the lungs;
2. provide lung expansion therapy and;
3. enhance delivery of aerosol therapy.

This "triple" mode device can provide aerosol therapy while alternating between CPEP for lung expansion and CHFO for airway clearance. Supplemental oxygen therapy may also be delivered when used with compressed oxygen.

The MN4000 has three therapy modes:

* CHFO (Continuous High Frequency Oscillation) - delivers aerosol therapy while providing oscillating pressure pulses to the airway
* CPEP (Continuous Positive Expiratory Pressure) - delivers aerosol therapy while providing continuous positive pressure to help hold open and expand the airways
* Aerosol - for delivery of aerosol only. In this mode, CHFO and CPEP are not available

After assessing baseline status, therapy with the MN4000 was introduced and incorporated into the daily home respiratory care treatment regimen for all patients.

Other airway clearance and/or lung expansion therapies were not to be performed during the three-month study period. The treatment regimen for other respiratory care modalities (e.g. aerosolized medications) was that which was prescribed by the patient's health care team in the routine standard care of each patient.

During the three-month follow-up period, adherence to the daily prescribed therapy regimen was assessed. Subjects/caregivers were asked to provide adherence information for each day during the 90-day study period.

Documentation of efficacy and safety Variables was completed by study staff at the time of occurrence, from review of the patient's medical records and from scores and rankings for questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of CF or MND
* Age ≥ 18 years
* Signed informed consent

Exclusion Criteria:

* Requirement for continuous mechanical ventilation
* Anticipated requirement for hospitalization within the next three months
* History of pneumothorax within past 6 months
* History of hemoptysis requiring embolization within past 12 months
* Inability to perform MN4000 therapy using a mouthpiece (e.g. inability to create adequate mouth seal)
* Inability to perform MN4000 therapy as directed
* Inability or unwillingness to complete study visits or provide follow-up data as required by the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa F Wolfe, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Home Based Airway Clearance With Metaneb: Patients with CF and MND who required regular home airway clearance therapy were enrolled to use the Metaneb device in the home setting.
Period: Overall Study
Arm/Group | Home Based Airway Clearance With Metaneb
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Home Based Airway Clearance With Metaneb in Patients With Cystic Fibrosis.: Patients with CF who required regular home airway clearance therapy were enrolled to use the Metaneb device in the home setting.
- Home Based Airway Clearance With Metaneb in Patients With Motor Neuron Disease.: Patients with MND who required regular home airway clearance therapy were enrolled to use the Metaneb device in the home setting.
- Total: Total of all reporting groups
Arm/Group | Home Based Airway Clearance With Metaneb in Patients With Cystic Fibrosis. | Home Based Airway Clearance With Metaneb in Patients With Motor Neuron Disease. | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.4 (4.34) | 65.2 (16.54) | 47.8 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 0 | 5 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Patient / Caregiver Satisfaction Scores
Description: The primary efficacy variable was patient and/or caregiver satisfaction with therapy, as evaluated using a Therapy Use Rating Questionnaire.
  The questionnaire was used to assess change in satisfaction or effectiveness on a variety of parameters.
  The satisfaction score was completed by the patient, if possible. Some of the patients in this study had Motor Neuron Disease. This disease can compromise the ability of the patient to interact and to respond to questions. In situations where patients could not respond, caregivers were asked to respond on their behalf.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Home Based Airway Clearance With Metaneb in Patients With Cystic Fibrosis. | Home Based Airway Clearance With Metaneb in Patients With Motor Neuron Disease.
Number analyzed (Participants) | 5 | 5
Participants
  Difficulty of Use (Day 30): Improved | 0 | 0
  Difficulty of Use (Day 30): Same | 4 | 4
  Difficulty of Use (Day 30): Worsened | 1 | 1
  Difficulty of Use (Day 30): Missing | 0 | 0
  Missed Treatment (Day 30): Improved | 2 | 2
  Missed Treatment (Day 30): Same | 2 | 2
  Missed Treatment (Day 30): Worsened | 1 | 1
  Missed Treatment (Day 30): Missing | 0 | 0
  Bring up sputum (Day 30): Improved | 1 | 4
  Bring up sputum (Day 30): Same | 3 | 0
  Bring up sputum (Day 30): Worsened | 1 | 1
  Bring up sputum (Day 30): Missing | 0 | 0
  Shortness of breath (Day 30): Improved | 0 | 2
  Shortness of breath (Day 30): Same | 2 | 0
  Shortness of breath (Day 30): Worsened | 1 | 1
  Shortness of breath (Day 30): Missing | 2 | 2
  Lungs stay healthy (Day 30): Improved | 0 | 3
  Lungs stay healthy (Day 30): Same | 4 | 2
  Lungs stay healthy (Day 30): Worsened | 1 | 0
  Lungs stay healthy (Day 30): Missing | 0 | 0
  Ability to perform tasks (Day 30): Improved | 1 | 1
  Ability to perform tasks (Day 30): Same | 2 | 2
  Ability to perform tasks (Day 30): Worsened | 2 | 2
  Ability to perform tasks (Day 30): Missing | 0 | 0
  Difficulty of Use (Day 90): Improved | 0 | 1
  Difficulty of Use (Day 90): Same | 3 | 3
  Difficulty of Use (Day 90): Worsened | 2 | 1
  Difficulty of Use (Day 90): Missing | 0 | 0
  Missed Treatment (Day 90): Improved | 3 | 1
  Missed Treatment (Day 90): Same | 1 | 3
  Missed Treatment (Day 90): Worsened | 1 | 1
  Missed Treatment (Day 90): Missing | 0 | 0
  Bring up sputum (Day 90): Improved | 1 | 4
  Bring up sputum (Day 90): Same | 2 | 0
  Bring up sputum (Day 90): Worsened | 2 | 1
  Bring up sputum (Day 90): Missing | 0 | 0
  Shortness of breath (Day 90): Improved | 1 | 2
  Shortness of breath (Day 90): Same | 1 | 0
  Shortness of breath (Day 90): Worsened | 1 | 1
  Shortness of breath (Day 90): Missing | 2 | 2
  Lungs stay healthy (Day 90): Improved | 0 | 3
  Lungs stay healthy (Day 90): Same | 3 | 1
  Lungs stay healthy (Day 90): Worsened | 2 | 1
  Lungs stay healthy (Day 90): Missing | 0 | 0
  Ability to perform tasks (Day 90): Improved | 0 | 2
  Ability to perform tasks (Day 90): Same | 2 | 2
  Ability to perform tasks (Day 90): Worsened | 3 | 1
  Ability to perform tasks (Day 90): Missing | 0 | 0

2. Primary Outcome: Patient / Caregiver Satisfaction Scores
Description: The Therapy Use Rating Questionnaire is an assessment of patient/caregiver satisfaction with the therapy and their subjective assessment of the benefit of the therapy.
  The questionnaire was used to assess change in satisfaction or effectiveness on a variety of parameters.
  The satisfaction score was completed by the patient, if possible. Some of the patients in this study had Motor Neuron Disease This disease can compromise the ability of the patient to interact and to respond to questions. In situations where patients could not respond, caregivers were asked to respond on their behalf.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Home Based Airway Clearance With Metaneb in Patients With Cystic Fibrosis. | Home Based Airway Clearance With Metaneb in Patients With Motor Neuron Disease.
Number analyzed (Participants) | 5 | 5
Participants
  Effective (Day 30): Much less | 0 | 0
  Effective (Day 30): Less | 1 | 0
  Effective (Day 30): Same | 2 | 2
  Effective (Day 30): More | 1 | 2
  Effective (Day 30): Much More | 1 | 1
  Easy to perform (Day 30): Much less | 1 | 0
  Easy to perform (Day 30): Less | 1 | 2
  Easy to perform (Day 30): Same | 1 | 1
  Easy to perform (Day 30): More | 1 | 1
  Easy to perform (Day 30): Much More | 1 | 1
  Like to continue MN4000 (Day 30): Much less | 1 | 0
  Like to continue MN4000 (Day 30): Less | 0 | 0
  Like to continue MN4000 (Day 30): Same | 0 | 0
  Like to continue MN4000 (Day 30): More | 1 | 0
  Like to continue MN4000 (Day 30): Much More | 3 | 5
  Effective (Day 90): Much less | 0 | 0
  Effective (Day 90): Less | 1 | 1
  Effective (Day 90): Same | 3 | 0
  Effective (Day 90): More | 0 | 1
  Effective (Day 90): Much More | 1 | 3
  Easy to perform (Day 90): Much less | 2 | 1
  Easy to perform (Day 90): Less | 2 | 0
  Easy to perform (Day 90): Same | 0 | 1
  Easy to perform (Day 90): More | 1 | 1
  Easy to perform (Day 90): Much More | 0 | 2
  Like to continue MN4000 (Day 90): Much less | 1 | 1
  Like to continue MN4000 (Day 90): Less | 1 | 0
  Like to continue MN4000 (Day 90): Same | 0 | 0
  Like to continue MN4000 (Day 90): More | 1 | 0
  Like to continue MN4000 (Day 90): Much More | 2 | 4

3. Secondary Outcome: Mean Percentage Adherence to Prescribed Treatment Regimen
Description: Adherence to the treatment regimen was calculated for each patient (number of minutes of therapy performed / number of minutes of therapy prescribed). The adherence percentage calculated for each study subject was then used to calculate the of Mean adherence to prescribed treatment regimen for the group or groups.
Time Frame: 90 days
Population: CF and MND population
Measure: Mean (Full Range); unit: Percentage of adherence to therapy
Groups:
- Patients With CF Who Required Home Based Airway Clearance With Metaneb: Patients with CF who required regular home airway clearance therapy were enrolled to use the Metaneb device in the home setting.
- Patients With MND Who Required Home Based Airway Clearance With Metaneb: Patients with MND who required regular home airway clearance therapy were enrolled to use the Metaneb device in the home setting.
Arm/Group | Patients With CF Who Required Home Based Airway Clearance With Metaneb | Patients With MND Who Required Home Based Airway Clearance With Metaneb
Number analyzed (Participants) | 5 | 5
Percentage of adherence to therapy | 97 [86 to 100] | 95 [89.7 to 99.5]

4. Secondary Outcome: ALS-Functional Rating Scale (ALS-FRS)
Description: MND patients only. The Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS) is an instrument for evaluating the functional status of patients with Amyotrophic Lateral Sclerosis. It can be used to monitor functional change in a patient over time.
  It contains 10 distinct measures:
  * Speech
  * Salivation
  * Swallowing
  * Handwriting
  * Cutting food and handling utensils (with or without gastrostomy)
  * Dressing and hygiene
  * Turning in bed and adjusting bed clothes
  * Walking
  * Breathing
  * Climbing stairs
  These 10 parameters are scored on a scale of 0-4, based on the patients' ability to perform tasks. The minimum score is 0 and maximum 40.The higher the score the more function is retained.
Time Frame: 90 days
Population: MND subpopulation
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Home Based Airway Clearance With Metaneb: ALS-Functional Rating Scale (ALS-FRS) of patients with Motor Neuron Disease
Arm/Group | Home Based Airway Clearance With Metaneb
Number analyzed (Participants) | 5
score on a scale
  Bulbar Sub-Score at Baseline | 10.8 (1.64)
  Bulbar Sub-Score after 30 days of therapy | 10.0 (3.39)
  Bulbar Sub-Score after 90 days of therapy | 10.4 (3.05)
  Respiratory Sub-score at baseline | 9.4 (1.52)
  Respiratory Sub-score after 30 days of therapy | 10.2 (1.10)
  Respiratory Sub-score after 90 days of therapy | 10.2 (1.10)
  Total Score at Baseline | 33.6 (6.84)
  Total Score after 30 days of therapy | 32.0 (5.29)
  Total Score after 90 days of therapy | 32.2 (5.07)

5. Secondary Outcome: Cystic Fibrosis Questionnaire - Revised (CFQ-R)
Description: CF patients only. The Cystic Fibrosis Questionnaire (CFQ) is a disease-specific instrument that measures health-related quality of life (HRQoL) for adolescents and adults with cystic fibrosis (CF) > or = 14 years, consisting of 44 items on 12 generic and disease-specific scales. It offers 5 distinct 4-point Likert scales (e.g., always/often/ sometime/never). Scores for each HRQoL domain; after recoding, each item is summed to generate a domain score and standardized. Scores range from 0 to 100, with higher scores indicating better health.
Time Frame: 90 days
Population: Cystic Fibrosis Questionnaire - Revised (CFQ-R) administered on the CF patient subpopulation
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Home Based Airway Clearance With Metaneb: Patients with CF who required regular home airway clearance therapy were enrolled to use the Metaneb device in the home setting.
Arm/Group | Home Based Airway Clearance With Metaneb
Number analyzed (Participants) | 5
Score on a scale
  Physical domain at baseline | 83.3 (19.54)
  Physical domain after 30 days of therapy | 78.3 (20.28)
  Physical domain after 90 days of therapy | 80.0 (17.78)
  Role domain at baseline | 80.0 (7.45)
  Role domain after 30 days of therapy | 90.0 (6.97)
  Role domain after 90 days of therapy | 86.7 (11.18)
  Vitality domain at baseline | 75.0 (16.67)
  Vitality domain after 30 days of therapy | 73.3 (6.97)
  Vitality domain after 90 days of therapy | 68.3 (13.69)
  Emotion domain at baseline | 89.3 (7.60)
  Emotion domain after 30 days of therapy | 81.3 (8.69)
  Emotion domain after 90 days of therapy | 86.7 (10.54)
  Social domain at baseline | 77.8 (14.70)
  Social domain after 30 days of therapy | 77.8 (13.61)
  Social domain after 90 days of therapy | 71.1 (13.83)
  Body domain at baseline | 97.8 (4.97)
  Body domain after 30 days of therapy | 91.1 (14.49)
  Body domain after 90 days of therapy | 91.1 (9.30)
  Eat domain at baseline | 97.8 (4.97)
  Eat domain after 30 days of therapy | 100.0 (0.00)
  Eat domain after 90 days of therapy | 100.0 (0.00)
  Treat domain at baseline | 55.6 (11.11)
  Treat domain after 30 days of therapy | 48.9 (9.94)
  Treat domain after 90 days of therapy | 46.7 (9.30)
  Health domain at baseline | 71.1 (6.09)
  Health domain after 30 days of therapy | 71.1 (6.09)
  Health domain after 90 days of therapy | 73.3 (14.91)
  Weight domain at baseline | 73.3 (36.51)
  Weight domain after 30 days of therapy | 100.0 (0.00)
  Weight domain after 90 days of therapy | 100.0 (0.00)
  Respiratory domain at baseline | 61.1 (23.90)
  Respiratory domain after 30 days of therapy | 61.1 (19.64)
  Respiratory domain after 90 days of therapy | 62.2 (10.69)
  Digestion domain at baseline | 84.4 (23.04)
  Digestion domain after 30 days of therapy | 93.3 (9.94)
  Digestion domain after 90 days of therapy | 91.1 (4.97)

6. Secondary Outcome: Number of Participants With Exacerbation of Pulmonary Disease
Description: Hospitalization and/or antibiotics for respiratory infection or complication. Exacerbations of pulmonary disease were defined as respiratory infections that resulted in the requirement for hospitalization and/or antibiotics to treat the respiratory infection or complication. Hospitalizations that are part of routine care (e.g. hospital admissions for annual "tune-up") or antibiotics that are part of the regular treatment regimen were not documented as exacerbations. Occurrence of exacerbation related hospitalization OR the necessity of a prescription for antibiotics qualify as worsening disease.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Home Based Airway Clearance With Metaneb
Number analyzed (Participants) | 10
Participants
  Exacerbation of pulmonary disease at baseline | 2
  Exacerbation that required antibiotics but not hospitalization at Day 30 | 1
  Exacerbations that required antibiotics at Day 90 | 3

7. Secondary Outcome: FEV1 (Actual)
Description: FEV1 is the actual volume measured in liters.
  Forced expiratory volume in one second (FEV1): The forced expiratory volume-one second is the total volume of air a patient exhales in the first second during maximal effort. Normal range is >80%. The patient takes a full breath in and exhale as hard and fast as they can. FEV1 refers to the volume of air that an individual can exhale during a forced breath in the first 1 second. Decreasing percentage is associated with worsening / severe disease
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Home Based Airway Clearance With Metaneb in Patients With Cystic Fibrosis. | Home Based Airway Clearance With Metaneb in Patients With Motor Neuron Disease.
Number analyzed (Participants) | 5 | 5
Liters
  FEV1 measure at baseline (Actual) | 1.8 (0.94) | 1.7 (0.54)
  FEV1 measure after 30 days of therapy (Actual) | 1.9 (1.05) | 1.6 (0.71)
  FEV1 measure after 90 days of therapy (Actual) | 1.9 (0.93) | 1.7 (0.73)

8. Secondary Outcome: FEV1 (% Predicted)
Description: FEV1 Percent Predicted (FEV1 % Predicted) is the actual volume exhaled in the first 1 second, divided by the "Normal" value for that actual value for a person of that age, gender, height and weight. A nomogram based on population norms provides a series of "Normal Values."
  FEV1: The forced expiratory volume-one second is the total volume of air a patient exhales in the first second during maximal effort. Normal range is >80%. Decreasing percentage is associated with worsening / severe disease
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: percentage of predicted normal
Arm/Group | Home Based Airway Clearance With Metaneb in Patients With Cystic Fibrosis. | Home Based Airway Clearance With Metaneb in Patients With Motor Neuron Disease.
Number analyzed (Participants) | 5 | 5
percentage of predicted normal
  FEV1 measure at baseline (% Predicted) | 55.2 (25.49) | 58.6 (19.49)
  FEV1 measure after 30 days of therapy (% Predicted) | 58.8 (27.81) | 57.8 (28.42)
  FEV1 measure after 90 days of therapy (% Predicted) | 60.4 (24.76) | 59.4 (27.67)

9. Secondary Outcome: FVC (Actual)
Description: FVC is the actual volume measured in liters.
  The functional vital capacity (FVC) is the total volume of air a patient exhales for the total duration of the test during maximal effort. Normal range is >80%. Decreasing percentage is associated with worsening / severe disease.
  FVC was only done in CF subjects because performance of the test requires intact respiratory muscle function. CF patients have intact respiratory muscle function and can therefore perform this maneuver. Patients with Motor Neuron Disease suffer from progressive weakness of all muscles including the respiratory muscles. The test results for FVC are affected muscle weakness and are therefore not a valid representation of their pulmonary function.
Time Frame: 90 days
Population: FVC and FEV1/FVC ratio are pulmonary function tests appropriate to assess lung function in patients with CF. These tests could not be physically performed by the patients in the MND population and thus these patients were not included in these analysis. For the MND population, SVC, SpO2, MIP, and PCF were performed instead of FVC and FEV1/FVC ratio. Hence, no data were collected from MND patients for this outcome measure.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Home Based Airway Clearance With Metaneb in Patients With Cystic Fibrosis.
Number analyzed (Participants) | 5
Liters
  FVC at baseline (Actual) | 2.6 (0.98)
  FVC after 30 days of therapy (Actual) | 2.6 (1.08)
  FVC after 90 days of therapy (Actual) | 2.7 (0.99)

10. Secondary Outcome: FVC (% Predicted)
Description: FVC Percent Predicted (FVC % Predicted) is the actual volume exhaled in the first 1 second, divided by the "Normal" value for that actual value for a person of that age, gender, height and weight. A nomogram based on population norms provides a series of "Normal Values."
  The functional vital capacity is the total volume of air a patient exhales for the total duration of the test during maximal effort. Normal range is >80%. Decreasing percentage is associated with worsening / severe disease.
  FVC was only done in CF subjects because performance of the test requires intact respiratory muscle function. CF patients have intact respiratory muscle function and can therefore perform this maneuver. Patients with Motor Neuron Disease suffer from progressive weakness of all muscles including the respiratory muscles. The test results for FVC are affected muscle weakness and are therefore not a valid representation of their pulmonary function.
Time Frame: 90 days
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage of predicted normal
Arm/Group | Home Based Airway Clearance With Metaneb in Patients With Cystic Fibrosis.
Number analyzed (Participants) | 5
percentage of predicted normal
  FVC at baseline (% Predicted) | 68.6 (22.09)
  FVC after 30 days of therapy (% Predicted) | 69.8 (23.19)
  FVC after 90 days of therapy (% Predicted) | 71.0 (21.30)

11. Secondary Outcome: FEV1/FVC Ratio
Description: The proportion of the FVC expired in one second Results are given in both actual values (litres, litres per second) and %predicted-the test result as a percent of the "predicted values" for the patients of similar characteristics. Results over 80% are considered normal.
  Patients with Motor Neuron Disease suffer from progressive weakness of all muscles including the respiratory muscles. The test results for FVC are affected muscle weakness and are therefore not a valid representation of their pulmonary function.
Time Frame: 90 days
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: FEV1/FVC ratio
Arm/Group | Home Based Airway Clearance With Metaneb
Number analyzed (Participants) | 5
FEV1/FVC ratio
  FEV1/FVC at baseline | 78.4 (19.78)
  FEV1/FVC after 30 days of therapy | 81.4 (18.42)
  FEV1/FVC after 90 days of therapy | 82.4 (14.54)

12. Secondary Outcome: SVC (Actual)
Description: Slow Vital Capacity (SVC) is the actual volume measured in liters.
  Slow Vital Capacity displays the volume of gas measured on a complete expiration after a maximal inspiration without forced or rapid effort. Useful measurement when FVC is reduced, and airway obstruction is present. Educed SVC is associated with worsening respiratory disease.
  Slow Vital Capacity provides the same measure as FVC - i.e. "Vital Capacity." It does not, however, require a "Forced expiratory maneuver (it requires a slow inspiration and slow expiration) and therefore is easier to achieve a valid result in patients with Motor Neuron Disease who suffer from progressive weakness of all muscles including the respiratory muscles.
Time Frame: 90 days
Population: FVC and FEV1/FVC ratio are pulmonary function tests appropriate to assess lung function in patients with CF. These tests could not be physically performed by the patients in the MND population and thus these patients were not included in these analysis. For the MND population, SVC, SpO2, MIP, and PCF were performed instead of FVC and FEV1/FVC ratio. Hence, no data were collected from CF patients for this outcome measure.
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- Home Based Airway Clearance With Metaneb: Patients with MND who required regular home airway clearance therapy were enrolled to use the Metaneb device in the home setting.
Arm/Group | Home Based Airway Clearance With Metaneb
Number analyzed (Participants) | 5
Liters
  SVC at baseline (Actual) | 2.1 (0.50)
  SVC after 30 days of therapy (Actual) | 2.2 (0.66)
  SVC after 90 days of therapy (Actual) | 2.1 (0.89)

13. Secondary Outcome: SVC (% Predicted)
Description: SVC Percent Predicted (SVC % Predicted) is the actual volume exhaled in the first 1 second, divided by the "Normal" value for that actual value for a person of that age, gender, height and weight. A nomogram based on population norms provides a series of "Normal Values."
  Slow Vital Capacity displays the volume of gas measured on a complete expiration after a maximal inspiration without forced or rapid effort. Useful measurement when FVC is reduced and airway obstruction is present. Educed SVC is associated with worsening respiratory disease.
  Slow Vital Capacity provides the same measure as FVC - i.e. "Vital Capacity." It does not, however, require a "Forced expiratory maneuver (it requires a slow inspiration and slow expiration) and therefore is easier to achieve a valid result in patients with Motor Neuron Disease who suffer from progressive weakness of all muscles including the respiratory muscles.
Time Frame: 90 days
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percentage of predicted normal
Arm/Group | Home Based Airway Clearance With Metaneb
Number analyzed (Participants) | 5
percentage of predicted normal
  SVC at baseline (% Predicted) | 55.2 (13.59)
  SVC after 30 days of therapy (% Predicted) | 58.2 (21.10)
  SVC after 90 days of therapy (% Predicted) | 54.6 (27.09)

14. Secondary Outcome: SpO2
Description: Standard pulmonary function measures (FEV1, FVC, and FEV1/FVC) are commonly followed in the clinical care of patients with CF.
  Standard pulmonary function measures (SVC, SpO2, MIP, and Peak Cough Flow) are commonly followed in the clinical care of patients with MND.
  SpO2 stands for peripheral capillary oxygen saturation, an estimate of the amount of oxygen in the blood. Low SpO2 is associated with worsening respiratory function.
Time Frame: 90 days
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percent of oxygen saturation
Arm/Group | Home Based Airway Clearance With Metaneb
Number analyzed (Participants) | 5
Percent of oxygen saturation
  SpO2 at baseline | 97.4 (0.89)
  SpO2 after 30 days of therapy | 96.8 (1.3)
  SpO2 after 90 days of therapy | 95.8 (1.64)

15. Secondary Outcome: Maximal Inspiratory Pressure (MIP)
Description: Standard pulmonary function measures (FEV1, FVC, and FEV1/FVC) are commonly followed in the clinical care of patients with CF.
  Standard pulmonary function measures (SVC, SpO2, MIP, and Peak Cough Flow) are commonly followed in the clinical care of patients with MND.
  Maximal inspiratory pressure (MIP) is a measure of the strength of inspiratory muscles, primarily the diaphragm, and allows for the assessment of ventilatory failure, restrictive lung disease and respiratory muscle strength. Reduction in MIP is asociated with worsening neuromuscular status and poor ability to cough.
Time Frame: 90 days
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Home Based Airway Clearance With Metaneb
Number analyzed (Participants) | 5
cmH2O
  MIP at baseline | -41.0 (21.24)
  MIP after 30 days of therapy | -35.6 (19.65)
  MIP at 90 days of therapy | -34.8 (15.32)

16. Secondary Outcome: PCF
Description: Standard pulmonary function measures (FEV1, FVC, and FEV1/FVC) are commonly followed in the clinical care of patients with CF.
  Standard pulmonary function measures (SVC, SpO2, MIP, and PCF) are commonly followed in the clinical care of patients with MND.
  The Peak Cough Flow (PCF) is the maximum air flow generated during a cough. Decreasing air flow generated is associated with weakening neuromuscular status and associated poor cough impulse
Time Frame: 90 days
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: liters per minute
Arm/Group | Home Based Airway Clearance With Metaneb
Number analyzed (Participants) | 5
liters per minute
  PCF at baseline | 344.0 (105.74)
  PCF after 30 days of therapy | 320.0 (152.81)
  PCF after 90 days of therapy: number analyzed (Participants) | 4
  PCF after 90 days of therapy | 280.0 (144.91)

ADVERSE EVENTS:
Time Frame: 90 days
Groups:
- Patients With CF Treated With Home Based Airway Clearance With Metaneb: Patients with CF who required regular home airway clearance therapy were enrolled to use the Metaneb device in the home setting.
- Patients With MND Treated With Home Based Airway Clearance With Metaneb: Patients with MND who required regular home airway clearance therapy were enrolled to use the Metaneb device in the home setting.
Arm/Group | Patients With CF Treated With Home Based Airway Clearance With Metaneb | Patients With MND Treated With Home Based Airway Clearance With Metaneb
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-05): https://cdn.clinicaltrials.gov/large-docs/77/NCT03797677/Prot_SAP_001.pdf